CLINICAL TRIAL: NCT00002199
Title: A Phase III Randomized Double-Blind, Multicenter Study to Evaluate the Safety and Efficacy of 3TC/ZDV/1592U89 and 3TC/ZDV/IDV in HIV-1 Infected Antiretroviral Therapy-Naive Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 238K; CNAA/B3005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Drug Resistance, Microbial; HIV Protease Inhibitors; Lamivudine; Indinavir; Genotype; Phenotype; Reverse Transcriptase Inhibitors; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; lamivudine, zidovudine drug combination; abacavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate

SUMMARY:
To compare the safety, tolerance, early antiviral activity, and durability of antiviral response of the lamivudine (3TC)/zidovudine (ZDV)/1592U89 arm versus the 3TC/ZDV/indinavir (IDV) arm. To determine the effect of the two arms on clinical efficacy as determined by the occurrence of new CDC, defined class B/C events, survival, medical resource utilization, and the development of plasma viral genotypic and phenotypic resistance.

DETAILED DESCRIPTION:
In this international study, 550 patients are randomized (225 per arm) to receive Combivir in combination with 1592U89 or indinavir. If after 16 weeks (and every 8 weeks thereafter until week 48) a patient has HIV-1 RNA >= 400 copies/ml (by PCR on two occasions >= 1 week and < 4 weeks apart), the patient has the option to switch to open-label therapy consisting of indinavir, 1592U89, and Combivir.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

GM-CSF, G-CSF, and erythropoietin.

Concurrent Treatment:

Allowed:

Local treatment for Kaposi's sarcoma.

Patients must have:

* HIV-1 infection documented by a licensed HIV-1 antibody ELISA and confirmed by Western blot detection of HIV-1 antibody or positive HIV-1 blood culture.
* CD4+ cell count >= 100 cells/mm3 within 14 days prior to study drug administration.
* HIV-1 RNA >= 10,000 copies/ml within 14 days prior to study drug administration.
* No active diagnosis of AIDS according to the 1993 Centers for Disease Control (CDC) AIDS surveillance definition (excluding CD4+ cell counts < 200 cells/mm3).
* Signed, informed consent from parent or legal guardian for patients under 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malabsorption syndrome or other gastrointestinal dysfunction that may interfere with drug absorption.
* Serious medical conditions such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction that would compromise the safety of the patient.

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapeutic agents.
* Agents with documented anti-HIV-1 activity in vitro.
* Foscarnet.
* Immunomodulating agents such as systemic corticosteroids, interleukins, thalidomide, or interferons.
* Terfenadine, astemizole, cisapride, triazolam, midazolam, and ergotamine/dihydroergotamine.

Concurrent Treatment:

Excluded:

* Radiation therapy.
* Other investigational treatments. NOTE:
* Treatments available through treatment IND or other expanded access programs are the exception and evaluated individually.

Patients with the following prior conditions are excluded:

History of relevant pancreatitis or hepatitis in the last 6 months.

Prior Medication:

Excluded:

* Cytotoxic chemotherapeutic agents within 30 days of study drug administration.
* Prior antiretroviral therapy.
* HIV vaccine dose within 90 days of study drug administration.
* Immunomodulating agents such as systemic corticosteroids, interleukins, or interferons within 30 days of study entry.

Prior Treatment:

Excluded:

Radiation therapy within 30 days of study drug administration.

Current alcohol or illicit drug use that may interfere with patient compliance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Med Ctr, Boston, Massachusetts, United States

REFERENCES:
- [Background] Staszewski S, Keiser P, Montaner J, Raffi F, Gathe J, Brotas V, Hicks C, Hammer SM, Cooper D, Johnson M, Tortell S, Cutrell A, Thorborn D, Isaacs R, Hetherington S, Steel H, Spreen W; CNAAB3005 International Study Team. Abacavir-lamivudine-zidovudine vs indinavir-lamivudine-zidovudine in antiretroviral-naive HIV-infected adults: A randomized equivalence trial. JAMA. 2001 Mar 7;285(9):1155-63. doi: 10.1001/jama.285.9.1155. PMID 11231744